CLINICAL TRIAL: NCT00152399
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled Trial To Study The Efficacy And The Safety Of The Early Administration Of Somatostatin (Ucb) 12 Mg/24 H IV Infusion And Two IV Boluses Of 250 Mcg During 72 Hours In The Treatment Of Subjects With Acute Severe Upper Gastrointestinal Bleeding (UGIB) With Suspicion Of Peptic Ulcer Bleeding [The PUB Study]
Brief Title: Study to Assess the Efficacy and Safety of Somatostatin in the Treatment of Acute Severe Upper Gastrointestinal Bleeding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9823
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Peptic Ulcer
Keywords: Peptic ulcer bleeding, upper intestinal bleeding, endoscopy, somatostatin
MeSH Terms: conditions — Peptic Ulcer; Peptic Ulcer Hemorrhage | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Somatostatin UCB (drug)

SUMMARY:
To assess the efficacy and safety of the early administration of somatostatin in infusion during 72 hours plus 2 boluses, compared to placebo in the control of acute severe UGIB with suspicion of PUB.

ELIGIBILITY:
Inclusion Criteria:

* Male or female non-cirrhotic patients at least 18 years old suspected to bleed from PU.
* Patients with haematemesis and/or hematochezia and/or melena which have been observed by a member of a clinical team (GP, hospital physician, nurse, ...).
* Either, documented signs of hypovolemia related to the current bleeding episode Or, occurrence of symptoms of hypovolemia

Exclusion Criteria:

* Treatment of the present bleeding episode with somatostatin or its analogues, vasoactive drugs, or endoscopic therapy.
* Any treatment with PPIs (IV or per os) within the last 48 hours preceding randomisation.
* Treatment (endotherapy or pharmacotherapy) for upper gastrointestinal ulcer bleeding in the last 30 days.
* Deficient haemostasis (platelets < 40 x 109/l, international normalised ratio of the prothrombin time > 1.5 (or prothrombin time < 70%), or activated partial thromboplastin time > 40 seconds (or according to the normal ranges validated, from local lab))
* Anticoagulant therapy (vitamin K antagonists or heparin including LMW heparins)
* Terminal stage illness in which endoscopy is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370
Dates: Start 2000-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of the early IV administration of somatostatin during 72 hours compared to placebo in the control of acute severe UGIB with suspicion of PUB by measuring the failure rate

SECONDARY OUTCOMES:
To evaluate the difference between somatostatin and placebo on the following variables; Type of failure; Time to failure(h) up to 72 hours; Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Kharkevitch, MD, Study Director — UCB Pharma
Locations (22):
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- France (5):
  - Angers
  - Bobigny
  - Créteil
  - Paris
  - Villejuif
- Greece (2):
  - Athens
  - Crete-Hellas
- Hungary (5):
  - Budapest
  - Debrecen
  - Győr
  - Kaposvár
  - Vác
- Poland (4):
  - Bydgoszcz
  - Krakow
  - Pruszków
  - Warsaw
- Spain (3):
  - Alicante
  - Barcelona
  - Madrid